CLINICAL TRIAL: NCT06390098
Title: A Phase 1, Open-Label, Positron Emission Tomography Study in Healthy Adult Subjects to Determine the Relationship Between Plasma Concentration and Brain Target Occupancy of ASN51 Following a Single Oral Dose
Brief Title: Positron Emission Tomography Study in Healthy Subjects to Determine the Relationship Between Plasma Concentration and Brain Target Occupancy of ASN51
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Asceneuron S.A. (Industry)
Collaborators: Hammersmith Medicines Research Invicro (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: ASN51-102
Record Dates: First submitted 2024-04-23; First posted 2024-04-30 (Actual); Results first posted 2025-05-08 (Actual); Last update posted 2025-05-08 (Actual); Status verified 2025-05

CONDITIONS: Healthy Participants

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ASN51 (Experimental): Participants received low, medium, and high doses of ASN51, orally on Day 1 of imaging sessions 2 and 3 before the PET scan during the study.
  Interventions: Drug: ASN51

INTERVENTIONS:
Drug: ASN51 — Oral

SUMMARY:
This is a phase 1, open-label, positron emission tomography (PET) study in healthy adult participants to determine the relationship between plasma concentration and brain target occupancy of ASN51 following a single oral dose.

ELIGIBILITY:
Inclusion Criteria:

* Healthy as determined by the Investigator, based on a medical evaluation including medical history physical examination, neurological examination, laboratory tests and cardiac monitoring. A participant with a clinical abnormality or laboratory parameters outside the reference range for the population being studied may be included only if, in the opinion of the Investigator, the finding is (a) unlikely to introduce additional risk to the participant, (b) will not interfere with study procedures or confound study results, and (c) is not otherwise exclusionary
* Men or women aged 25-55 years, inclusive (age range was selected on grounds of radiation burden).
* Women of child-bearing potential (WOCBP) with partners of child-bearing potential must agree to use highly effective contraception from at least 28 days before first tracer dosing through 30 days after last dose of study medication. All WOCBP must have a negative pregnancy test result before administration of test article. Vasectomized partner is also an accepted a highly effective birth control method provided that partner is the sole sexual partner of the WOCBP trial participant and that the vasectomized partner has received medical assessment of the surgical success.
* WOCBP must be postmenopausal (the last menstrual period was at least 12 months ago, and follicle-stimulating hormone at screening confirms postmenopausal status, or have no uterus, ovaries, or fallopian tubes). Women who are surgically sterile must provide documentation of the procedure by an operative report or by ultrasound.
* Non-sterilized male participants who are not abstinent and intend to be sexually active with a female partner of childbearing potential must use a male condom plus spermicide from 1 day prior to the first tracer administration throughout the total duration of the treatment period and 90 days after the last dose of study drug. Periodic abstinence, the rhythm method, and the withdrawal method are not acceptable methods of contraception. Male participants should refrain from sperm donation throughout this period.
* Body weight > 50.0 kilograms (kg) for men and > 45.0 kg for women and Body Mass Index within the range 18.5-30.0 kilograms per square meter (kg/m^2) (inclusive).
* Participants must understand the nature of the study and must provide signed and dated written informed consent in accordance with local regulations before the conduct of any study-related procedures.
* Participants must be, in the opinion of the Investigator, able to participate in all scheduled evaluations, likely to complete all required tests, and likely to be compliant.
* Participants must be fluent in the local language.
* Participants must agree not to post any personal medical data related to the study or information related to the study on any website or social media site (e.g., Facebook, Twitter, etc.) until the trial has completed.

Exclusion Criteria:

* A positive urine drug screen/alcohol test at Screening or Day -1.
* Any history of psychiatric disorders, including substance use disorders, according to the Diagnostic and Statistical Manual of Mental Disorders, 5th Edition (DSM-5) criteria.
* A diagnosis of intellectual disability (intellectual developmental disorder) or mental retardation.
* Significant suicide risk as assessed by the Columbia Suicide severity Rating Scale (C-SSRS)
* A positive Hepatitis B surface antigen or positive Hepatitis C antibody result at Screening.
* A positive test for human immunodeficiency virus (HIV) antibody at Screening.
* Alanine aminotransferase or aspartate aminotransferase levels greater than 1.5 times the upper limit of normal (ULN) at Screening or between Screening and first dose of tracer.
* Frequently used any tobacco-containing (e.g., cigar, cigarette, or snuff) or nicotine-containing product (e.g., nicotine chewing gum, nicotine plasters, or other product used for smoking cessation) within 3 months prior to first dose of tracer. Frequent use is defined as 3 or more days per week. Use of any tobacco- or nicotine-containing product is prohibited within 1 week of first dose of tracer.
* History of regular alcohol consumption within 12 months of the study defined as an average weekly intake of >21 alcoholic units/week for men or >14 alcoholic units/week for women.
* Regularly consumed (e.g., more days than not) excessive quantities of xanthine-containing beverages (e.g., more than five cups of coffee or the equivalent per day) within 30 days prior to Screening or between Screening and first dose of tracer.
* Received or used an investigational product (including placebo) or device within the following time period prior to the first tracer dosing day in the current study: 90 days, 5 half-lives or twice the duration of the biological effect of the investigational product (whichever is longer).
* Use of prescription or non-prescription drugs, vitamins, herbal, and dietary supplements (including St John's Wort) within 7 days (or 28 days if the drug is a potential hepatic enzyme inducer) or 5 half-lives (whichever is longer) prior to the first dose of study tracer medication, unless in the opinion of the Investigator and Medical Monitor, the medication will not interfere with the study procedures or compromise Participant safety.
* History of clinically significant sensitivity to any of the study medications, or components thereof or a history of drug or other allergy that, in the opinion of the Investigator or Medical Monitor, contraindicates their participation.
* Loss of more than 400 milliliters (mL) of blood within 3 months prior to first dose of tracer, i.e., blood donor.
* A positive serum pregnancy test or lactation.
* A history or presence of any disease, condition, or surgery likely to affect drug absorption, distribution, metabolism, or excretion. Participants with a history of cholecystectomy should be excluded.
* A history or presence of a clinically significant hepatic, renal, gastrointestinal, cardiovascular, endocrine, pulmonary, ophthalmologic, immunologic, hematologic, dermatologic, or neurologic abnormality.
* A clinically significant abnormality on physical examination, neurological examination, electrocardiogram (ECG), or laboratory evaluations at screen or between screen and first tracer dose administration.
* A corrected QT(total time from ventricular depolarization to complete repolarization) interval measurement corrected according to the Fridericia rule (QTcF) > 450 milliseconds (msec) for males and 470 msec for females during controlled rest at screen or between screen and first tracer dose administration, or family history of long QT syndrome.
* Any clinically significant abnormalities in rhythm, conduction, or morphology of the resting ECG and any abnormalities in the 12-lead ECG that, in the judgement of the Investigator or Medical Monitor, may interfere with the interpretation of QTc interval changes, including abnormal ST-T-wave morphology or left ventricular hypertrophy.
* PR (PQ) interval shortening < 120 msec (PR < 120 msec but > 110 msec is acceptable if there is no evidence of ventricular pre-excitation).
* PR (PQ) interval prolongation (>220 msec), intermittent second- (Wenckebach block while asleep or in deep rest is not exclusionary) or third-degree AV block.
* Persistent or intermittent complete bundle branch block (BBB), incomplete bundle branch block (IBBB), or intraventricular conduction delay (IVCD) with QRS > 120 msec.
* A clinically significant vital signs abnormality at screening This includes, but is not limited to, 3 measurements (each 5 minutes apart) in the seated position: (a) systolic blood pressure < 90 or >140 millimeters of mercury (mmHg), (b) diastolic blood pressure <50 or > 95 mmHg, or (c) heart rate < 45 or >100 beats per minute. The average of the 3 measurements should be used to assess eligibility at screening.
* Significant (> 10%) weight loss or gain within 30 days prior to Screening and first tracer dose administration.
* A history of seizure. History of a single benign febrile convulsion of childhood is permitted.
* A history of head trauma, including closed head injury with loss of consciousness.
* A history of symptomatic orthostatic hypotension (i.e., postural syncope).
* A history of neuroleptic malignant syndrome.
* A history of chronic urinary tract infections.
* The participant is, in the opinion of the Investigator or Medical Monitor, unlikely to comply with the protocol or is unsuitable for any reason.
* Currently employed by Asceneuron SA or by a clinical trial site participating in this study, or a first-degree relative of an Asceneuron SA employee or of an employee at a participating clinical trial site.
* Unsatisfactory venous access
* Significant exposure to ionizing radiation as part of research within the previous 12 months prior to first tracer dose administration.
* Unsuitable or unwilling to undergo the imaging procedures, as determined by an magnetic resonance imaging (MRI) safety questionnaire. Reasons for exclusion include but are not limited to presence of a cardiac pacemaker or other implanted electronic device; ferromagnetic metal foreign bodies, intracranial aneurysm clips or other metallic objects; non-MRI compatible heart valves; inner ear implants; or a history of claustrophobia.
* Significant structural brain abnormality, as determined by MRI.
* Contraindication for arterial cannulation: Allen's test indicating potential risk in placement of the arterial cannula.
* Participants with a COVID-19 vaccination within two weeks of screening or due to receive second dose of COVID-19 vaccine while participating in the study.

Ages: 25 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 3 (Actual)
Dates: Start 2021-08-09 (Actual); Primary Completion 2021-10-12 (Actual); Study Completion 2021-10-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Hammersmith, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Not expected to be made available

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at an investigative site in United Kingdom from 09 August 2021 to 12 October 2021.
Groups:
- ASN51: All participants received low, medium, and high doses of ASN51 (as assigned according to the protocol), orally on Day 1 of imaging sessions 2 and 3 before the positron emission tomography (PET) scan during the study.
Period: Overall Study
Arm/Group | ASN51
Started | 3
Completed | 3
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: All treated set included all participants who received at least one dose of study drug.
Arm/Group | ASN51
Number analyzed (Participants) | 3
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.3 (4.93)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 3
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 3
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Regional Total Volume of Distribution (VT) of [18F]-IMA601 in Frontal Lobe at Each Brain Scan
Description: Regional VT of [18F]-IMA601 in frontal lobe at each brain scan was measured with a PET scan. Participants received an intravenous (IV) dose of the radiolabelled tracer, [18F]-IMA601, at the start of each PET scan. Participant wise data was reported for this outcome measure.
Time Frame: PET Scan 1 (Baseline), PET Scan 2 (6 hours post-dose [for participant 1] and 31 hours post-dose for [participants 2 and 3] on Day 1), PET Scan 3 (48 hours post-dose on Day 1) after final ASN51 dose
Population: PET population included all participants who received study medication, had a baseline PET scan, at least one post-baseline PET scan, and a pharmacokinetic (PK) result immediately preceding PET scan. Here, "number analyzed" signifies specific participant evaluated in respective arm at a specified timepoint.
Measure: Number; unit: milliliters/cubic centimeter (mL/cm^3)
Groups:
- All Participants: Participants participated in imaging session 1 (Baseline) of PET scan before dosing during the study.
- ASN51 Low Dose: Participants received low dose of ASN51, orally on Day 1 of imaging sessions 2 and 3 before the PET scan during the study.
- ASN51 Medium Dose: Participants received medium dose of ASN51, orally on Day 1 of imaging sessions 2 and 3 before the PET scan during the study.
- ASN51 High Dose: Participants received high dose of ASN51, orally on Day 1 of imaging sessions 2 and 3 before the PET scan during the study.
Arm/Group | All Participants | ASN51 Low Dose | ASN51 Medium Dose | ASN51 High Dose
Number analyzed (Participants) | 3 | 3 | 1 | 1
milliliters/cubic centimeter (mL/cm^3)
  Participant 1, PET Scan 1, Baseline: number analyzed (Participants) | 1 | 0 | 0 | 0
  Participant 1, PET Scan 1, Baseline | 14.09 |  |  |
  Participant 1, PET Scan 2, 6 hours post-dose, Day 1: number analyzed (Participants) | 0 | 0 | 0 | 1
  Participant 1, PET Scan 2, 6 hours post-dose, Day 1 |  |  |  | 1.82
  Participant 1, PET Scan 3, 48 hours post-dose, Day 1: number analyzed (Participants) | 0 | 1 | 0 | 0
  Participant 1, PET Scan 3, 48 hours post-dose, Day 1 |  | 4.76 |  |
  Participant 2, PET Scan 1, Baseline: number analyzed (Participants) | 1 | 0 | 0 | 0
  Participant 2, PET Scan 1, Baseline | 16.08 |  |  |
  Participant 2, PET Scan 2, 31 hours post-dose, Day 1: number analyzed (Participants) | 0 | 1 | 0 | 0
  Participant 2, PET Scan 2, 31 hours post-dose, Day 1 |  | 3.90 |  |
  Participant 2, PET Scan 3, 48 hours post-dose, Day 1: number analyzed (Participants) | 0 | 1 | 0 | 0
  Participant 2, PET Scan 3, 48 hours post-dose, Day 1 |  | 4.55 |  |
  Participant 3, PET Scan 1, Baseline: number analyzed (Participants) | 1 | 0 | 0 | 0
  Participant 3, PET Scan 1, Baseline | 16.38 |  |  |
  Participant 3, PET Scan 2, 31 hours post-dose, Day 1: number analyzed (Participants) | 0 | 0 | 1 | 0
  Participant 3, PET Scan 2, 31 hours post-dose, Day 1 |  |  | 3.86 |
  Participant 3, PET Scan 3, 48 hours post-dose, Day 1: number analyzed (Participants) | 0 | 1 | 0 | 0
  Participant 3, PET Scan 3, 48 hours post-dose, Day 1 |  | 5.78 |  |

2. Primary Outcome: Regional VT of [18F]-IMA601 in Anterior Cingulate at Each Brain Scan
Description: Regional VT of [18F]-IMA601 in anterior cingulate at each brain scan was measured with a PET scan. Participants received an IV dose of the radiolabelled tracer, [18F]-IMA601, at the start of each PET scan. Participant wise data was reported for this outcome measure.
Time Frame: as for outcome 1
Population: PET population included all participants who received study medication, had a baseline PET scan, at least one post-baseline PET scan, and a PK result immediately preceding PET scan. Here, "number analyzed" signifies specific participant evaluated in respective arm at a specified timepoint.
Measure: Number; unit: mL/cm^3
Arm/Group | All Participants | ASN51 Low Dose | ASN51 Medium Dose | ASN51 High Dose
Number analyzed (Participants) | 3 | 3 | 1 | 1
mL/cm^3
  Participant 1, PET Scan 1, Baseline: number analyzed (Participants) | 1 | 0 | 0 | 0
  Participant 1, PET Scan 1, Baseline | 16.35 |  |  |
  Participant 1, PET Scan 2, 6 hours post-dose, Day 1: number analyzed (Participants) | 0 | 0 | 0 | 1
  Participant 1, PET Scan 2, 6 hours post-dose, Day 1 |  |  |  | 1.85
  Participant 1, PET Scan 3, 48 hours post-dose: number analyzed (Participants) | 0 | 1 | 0 | 0
  Participant 1, PET Scan 3, 48 hours post-dose |  | 5.41 |  |
  Participant 2, PET Scan 1, Baseline: number analyzed (Participants) | 1 | 0 | 0 | 0
  Participant 2, PET Scan 1, Baseline | 19.34 |  |  |
  Participant 2, PET Scan 2, 31 hours post-dose, Day 1: number analyzed (Participants) | 0 | 1 | 0 | 0
  Participant 2, PET Scan 2, 31 hours post-dose, Day 1 |  | 4.28 |  |
  Participant 2, PET Scan 3, 48 hours post-dose, Day 1: number analyzed (Participants) | 0 | 1 | 0 | 0
  Participant 2, PET Scan 3, 48 hours post-dose, Day 1 |  | 5.13 |  |
  Participant 3, PET Scan 1, Baseline: number analyzed (Participants) | 1 | 0 | 0 | 0
  Participant 3, PET Scan 1, Baseline | 19.89 |  |  |
  Participant 3, PET Scan 2, 31 hours post-dose, Day 1: number analyzed (Participants) | 0 | 0 | 1 | 0
  Participant 3, PET Scan 2, 31 hours post-dose, Day 1 |  |  | 4.21 |
  Participant 3, PET Scan 3, 48 hours post-dose, Day 1: number analyzed (Participants) | 0 | 1 | 0 | 0
  Participant 3, PET Scan 3, 48 hours post-dose, Day 1 |  | 6.70 |  |

3. Primary Outcome: Regional VT of [18F]-IMA601 in Caudate at Each Brain Scan
Description: Regional VT of [18F]-IMA601 in the caudate at each brain scan was measured with a PET scan. Participants received an IV dose of the radiolabelled tracer, [18F]-IMA601, at the start of each PET scan. Participant wise data was reported for this outcome measure.
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Number; unit: mL/cm^3
Arm/Group | All Participants | ASN51 Low Dose | ASN51 Medium Dose | ASN51 High Dose
Number analyzed (Participants) | 3 | 3 | 1 | 1
mL/cm^3
  Participant 1, PET Scan 1, Baseline: number analyzed (Participants) | 1 | 0 | 0 | 0
  Participant 1, PET Scan 1, Baseline | 10.20 |  |  |
  Participant 1, PET Scan 2, 6 hours post-dose, Day 1: number analyzed (Participants) | 0 | 0 | 0 | 1
  Participant 1, PET Scan 2, 6 hours post-dose, Day 1 |  |  |  | 1.23
  Participant 1, PET Scan 3, 48 hours post-dose, Day 1: number analyzed (Participants) | 0 | 1 | 0 | 0
  Participant 1, PET Scan 3, 48 hours post-dose, Day 1 |  | 3.21 |  |
  Participant 2, PET Scan 1, Baseline: number analyzed (Participants) | 1 | 0 | 0 | 0
  Participant 2, PET Scan 1, Baseline | 13.74 |  |  |
  Participant 2, PET Scan 2, 31 hours post-dose, Day 1: number analyzed (Participants) | 0 | 1 | 0 | 0
  Participant 2, PET Scan 2, 31 hours post-dose, Day 1 |  | 3.19 |  |
  Participant 2, PET Scan 3, 48 hours post-dose, Day 1: number analyzed (Participants) | 0 | 1 | 0 | 0
  Participant 2, PET Scan 3, 48 hours post-dose, Day 1 |  | 3.89 |  |
  Participant 3, PET Scan 1, Baseline: number analyzed (Participants) | 1 | 0 | 0 | 0
  Participant 3, PET Scan 1, Baseline | 14.70 |  |  |
  Participant 3, PET Scan 2, 31 hours post-dose, Day 1: number analyzed (Participants) | 0 | 0 | 1 | 0
  Participant 3, PET Scan 2, 31 hours post-dose, Day 1 |  |  | 3.31 |
  Participant 3, PET Scan 3, 48 hours post-dose, Day 1: number analyzed (Participants) | 0 | 1 | 0 | 0
  Participant 3, PET Scan 3, 48 hours post-dose, Day 1 |  | 4.86 |  |

4. Primary Outcome: Regional VT of [18F]-IMA601 in Putamen at Each Brain Scan
Description: Regional VT of [18F]-IMA601 in putamen at each brain scan was measured with a PET scan. Participants received an IV dose of the radiolabelled tracer, [18F]-IMA601, at the start of each PET scan. Participant wise data was reported for this outcome measure.
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Number; unit: mL/cm^3
Arm/Group | All Participants | ASN51 Low Dose | ASN51 Medium Dose | ASN51 High Dose
Number analyzed (Participants) | 3 | 3 | 1 | 1
mL/cm^3
  Participant 1, PET Scan 1, Baseline: number analyzed (Participants) | 1 | 0 | 0 | 0
  Participant 1, PET Scan 1, Baseline | 15.38 |  |  |
  Participant 1, PET Scan 2, 6 hours post-dose, Day 1: number analyzed (Participants) | 0 | 0 | 0 | 1
  Participant 1, PET Scan 2, 6 hours post-dose, Day 1 |  |  |  | 1.98
  Participant 1, PET Scan 3, 48 hours post-dose, Day 1: number analyzed (Participants) | 0 | 1 | 0 | 0
  Participant 1, PET Scan 3, 48 hours post-dose, Day 1 |  | 5.41 |  |
  Participant 2, PET Scan 1, Baseline: number analyzed (Participants) | 1 | 0 | 0 | 0
  Participant 2, PET Scan 1, Baseline | 19.07 |  |  |
  Participant 2, PET Scan 2, 31 hours post-dose, Day 1: number analyzed (Participants) | 0 | 1 | 0 | 0
  Participant 2, PET Scan 2, 31 hours post-dose, Day 1 |  | 4.37 |  |
  Participant 2, PET Scan 3, 48 hours post-dose, Day 1: number analyzed (Participants) | 0 | 1 | 0 | 0
  Participant 2, PET Scan 3, 48 hours post-dose, Day 1 |  | 5.22 |  |
  Participant 3, PET Scan 1, Baseline: number analyzed (Participants) | 1 | 0 | 0 | 0
  Participant 3, PET Scan 1, Baseline | 19.32 |  |  |
  Participant 3, PET Scan 2, 31 hours post-dose, Day 1: number analyzed (Participants) | 0 | 0 | 1 | 0
  Participant 3, PET Scan 2, 31 hours post-dose, Day 1 |  |  | 4.39 |
  Participant 3, PET Scan 3, 48 hours post-dose, Day 1: number analyzed (Participants) | 0 | 1 | 0 | 0
  Participant 3, PET Scan 3, 48 hours post-dose, Day 1 |  | 6.57 |  |

5. Primary Outcome: Regional VT of [18F]-IMA601 in Accumbens at Each Brain Scan
Description: Regional VT of [18F]-IMA601 in accumbens at each brain scan was measured with a PET scan. Participants received an IV dose of the radiolabelled tracer, [18F]-IMA601, at the start of each PET scan. Participant wise data was reported for this outcome measure.
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Number; unit: mL/cm^3
Arm/Group | All Participants | ASN51 Low Dose | ASN51 Medium Dose | ASN51 High Dose
Number analyzed (Participants) | 3 | 3 | 1 | 1
mL/cm^3
  Participant 1, PET Scan 1, Baseline: number analyzed (Participants) | 1 | 0 | 0 | 0
  Participant 1, PET Scan 1, Baseline | 15.82 |  |  |
  Participant 1, PET Scan 2, 6 hours post-dose, Day 1: number analyzed (Participants) | 0 | 0 | 0 | 1
  Participant 1, PET Scan 2, 6 hours post-dose, Day 1 |  |  |  | 1.69
  Participant 1, PET Scan 3, 48 hours post-dose, Day 1: number analyzed (Participants) | 0 | 1 | 0 | 0
  Participant 1, PET Scan 3, 48 hours post-dose, Day 1 |  | 5.43 |  |
  Participant 2, PET Scan 1, Baseline: number analyzed (Participants) | 1 | 0 | 0 | 0
  Participant 2, PET Scan 1, Baseline | 21.14 |  |  |
  Participant 2, PET Scan 2, 31 hours post-dose, Day 1: number analyzed (Participants) | 0 | 1 | 0 | 0
  Participant 2, PET Scan 2, 31 hours post-dose, Day 1 |  | 4.42 |  |
  Participant 2, PET Scan 3, 48 hours post-dose, Day 1: number analyzed (Participants) | 0 | 1 | 0 | 0
  Participant 2, PET Scan 3, 48 hours post-dose, Day 1 |  | 5.36 |  |
  Participant 3, PET Scan 1, Baseline: number analyzed (Participants) | 1 | 0 | 0 | 0
  Participant 3, PET Scan 1, Baseline | 21.80 |  |  |
  Participant 3, PET Scan 2, 31 hours post-dose, Day 1: number analyzed (Participants) | 0 | 0 | 1 | 0
  Participant 3, PET Scan 2, 31 hours post-dose, Day 1 |  |  | 4.28 |
  Participant 3, PET Scan 3, 48 hours post-dose, Day 1: number analyzed (Participants) | 0 | 1 | 0 | 0
  Participant 3, PET Scan 3, 48 hours post-dose, Day 1 |  | 6.71 |  |

6. Primary Outcome: Regional VT of [18F]-IMA601 in Amygdala at Each Brain Scan
Description: Regional VT of [18F]-IMA601 in amygdala at each brain scan was measured with a PET scan. Participants received an IV dose of the radiolabelled tracer, [18F]-IMA601, at the start of each PET scan. Participant wise data was reported for this outcome measure.
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Number; unit: mL/cm^3
Arm/Group | All Participants | ASN51 Low Dose | ASN51 Medium Dose | ASN51 High Dose
Number analyzed (Participants) | 3 | 3 | 1 | 1
mL/cm^3
  Participant 1, PET Scan 1, Baseline: number analyzed (Participants) | 1 | 0 | 0 | 0
  Participant 1, PET Scan 1, Baseline | 16.40 |  |  |
  Participant 1, PET Scan 2, 6 hours post-dose, Day 1: number analyzed (Participants) | 0 | 0 | 0 | 1
  Participant 1, PET Scan 2, 6 hours post-dose, Day 1 |  |  |  | 1.90
  Participant 1, PET Scan 3, 48 hours post-dose, Day 1: number analyzed (Participants) | 0 | 1 | 0 | 0
  Participant 1, PET Scan 3, 48 hours post-dose, Day 1 |  | 6.36 |  |
  Participant 2, PET Scan 1, Baseline: number analyzed (Participants) | 1 | 0 | 0 | 0
  Participant 2, PET Scan 1, Baseline | 22.30 |  |  |
  Participant 2, PET Scan 2, 31 hours post-dose, Day 1: number analyzed (Participants) | 0 | 1 | 0 | 0
  Participant 2, PET Scan 2, 31 hours post-dose, Day 1 |  | 4.76 |  |
  Participant 2, PET Scan 3, 48 hours post-dose, Day 1: number analyzed (Participants) | 0 | 1 | 0 | 0
  Participant 2, PET Scan 3, 48 hours post-dose, Day 1 |  | 6.00 |  |
  Participant 3, PET Scan 1, Baseline: number analyzed (Participants) | 1 | 0 | 0 | 0
  Participant 3, PET Scan 1, Baseline | 22.18 |  |  |
  Participant 3, PET Scan 2, 31 hours post-dose, Day 1: number analyzed (Participants) | 0 | 0 | 1 | 0
  Participant 3, PET Scan 2, 31 hours post-dose, Day 1 |  |  | 4.49 |
  Participant 3, PET Scan 3, 48 hours post-dose, Day 1: number analyzed (Participants) | 0 | 1 | 0 | 0
  Participant 3, PET Scan 3, 48 hours post-dose, Day 1 |  | 7.26 |  |

7. Primary Outcome: Regional VT of [18F]-IMA601 in Cerebral White Matter at Each Brain Scan
Description: Regional VT of [18F]-IMA601 in cerebral white matter at each brain scan was measured with a PET scan. Participants received an IV dose of the radiolabelled tracer, [18F]-IMA601, at the start of each PET scan. Participant wise data was reported for this outcome measure.
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Number; unit: mL/cm^3
Arm/Group | All Participants | ASN51 Low Dose | ASN51 Medium Dose | ASN51 High Dose
Number analyzed (Participants) | 3 | 3 | 1 | 1
mL/cm^3
  Participant 1, PET Scan 1, Baseline: number analyzed (Participants) | 1 | 0 | 0 | 0
  Participant 1, PET Scan 1, Baseline | 10.87 |  |  |
  Participant 1, PET Scan 2, 6 hours post-dose, Day 1: number analyzed (Participants) | 0 | 0 | 0 | 1
  Participant 1, PET Scan 2, 6 hours post-dose, Day 1 |  |  |  | 1.72
  Participant 1, PET Scan 3, 48 hours post-dose, Day 1: number analyzed (Participants) | 0 | 1 | 0 | 0
  Participant 1, PET Scan 3, 48 hours post-dose, Day 1 |  | 3.86 |  |
  Participant 2, PET Scan 1, Baseline: number analyzed (Participants) | 1 | 0 | 0 | 0
  Participant 2, PET Scan 1, Baseline | 12.72 |  |  |
  Participant 2, PET Scan 2, 31 hours post-dose, Day 1: number analyzed (Participants) | 0 | 1 | 0 | 0
  Participant 2, PET Scan 2, 31 hours post-dose, Day 1 |  | 3.32 |  |
  Participant 2, PET Scan 3, 48 hours post-dose: number analyzed (Participants) | 0 | 1 | 0 | 0
  Participant 2, PET Scan 3, 48 hours post-dose |  | 3.80 |  |
  Participant 3, PET Scan 1, Baseline: number analyzed (Participants) | 1 | 0 | 0 | 0
  Participant 3, PET Scan 1, Baseline | 13.49 |  |  |
  Participant 3, PET Scan 2, 31 hours post-dose, Day 1: number analyzed (Participants) | 0 | 0 | 1 | 0
  Participant 3, PET Scan 2, 31 hours post-dose, Day 1 |  |  | 3.58 |
  Participant 3, PET Scan 3, 48 hours post-dose, Day 1: number analyzed (Participants) | 0 | 1 | 0 | 0
  Participant 3, PET Scan 3, 48 hours post-dose, Day 1 |  | 4.97 |  |

8. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs) and Serious TEAEs
Description: An adverse event (AE) is any untoward medical occurrence associated with the use of a drug in humans, whether or not considered drug related. TEAE is defined as an AE that emerges during treatment (having been absent before treatment) or that worsens after treatment. Serious TEAE is defined as an event that results in death, is considered life threatening, requires in-patient hospitalization or prolongation of existing hospitalization, results in persistent/significant disability/incapacity, results in a congenital anomaly/birth defect; or other medially important serious medical event.
Time Frame: Up to approximately 2.1 months
Population: Safety analysis set included all participants from the all-treated set who had at least one safety assessment post-baseline.
Measure: Count of Participants; unit: Participants
Arm/Group | All Participants | ASN51 Low Dose | ASN51 Medium Dose | ASN51 High Dose
Number analyzed (Participants) | 3 | 3 | 1 | 1
Participants
  Participants with TEAEs | 2 | 0 | 1 | 0
  Participants with Serious TEAEs | 0 | 0 | 0 | 0

9. Secondary Outcome: Number of Participants With Serious TEAEs up to 4 Weeks After Last Administration
Description: An AE is any untoward medical occurrence associated with the use of a drug in humans, whether or not considered drug related. Serious TEAE is defined as an event that results in death, is considered life threatening, requires in-patient hospitalization or prolongation of existing hospitalization, results in persistent/significant disability/incapacity, results in a congenital anomaly/birth defect; or other medially important serious medical event.
Time Frame: Up to 4 weeks
Population: as for outcome 8
Measure: Count of Participants; unit: Participants
Arm/Group | All Participants | ASN51 Low Dose | ASN51 Medium Dose | ASN51 High Dose
Number analyzed (Participants) | 3 | 3 | 1 | 1
Participants | 0 | 0 | 0 | 0

10. Secondary Outcome: Number of Participants With Clinically Significant Abnormalities in Laboratory Parameters
Description: Laboratory tests including hematology, biochemistry, coagulation, serology, pregnancy and follicle stimulating hormone (FSH) test (only for females), and urinalysis were performed. Number of participants with clinically significant abnormalities in laboratory parameters were reported. Clinical significance was determined by the investigator.
Time Frame: Up to approximately 2.1 months
Population: as for outcome 8
Measure: Count of Participants; unit: Participants
Arm/Group | All Participants | ASN51 Low Dose | ASN51 Medium Dose | ASN51 High Dose
Number analyzed (Participants) | 3 | 3 | 1 | 1
Participants | 0 | 0 | 0 | 0

11. Secondary Outcome: Number of Participants With Clinically Significant Changes in Vital Signs
Description: Vital signs including seated systolic blood pressure, seated diastolic blood pressure, seated heart rate, respiratory rate, and tympanic temperature were assessed. Number of participants with clinically significant changes in vital signs were reported. Clinical significance was determined by the investigator.
Time Frame: Up to approximately 2.1 months
Population: as for outcome 8
Measure: Count of Participants; unit: Participants
Arm/Group | All Participants | ASN51 Low Dose | ASN51 Medium Dose | ASN51 High Dose
Number analyzed (Participants) | 3 | 3 | 1 | 1
Participants | 0 | 0 | 0 | 0

12. Secondary Outcome: Number of Participants With Clinically Significant Abnormal Electrocardiogram (ECG) Findings
Description: ECG parameters including Ventricular rate, QRS complex of the ECG reflects the rapid depolarization of the right and left ventricles (QRS) interval, portion of the ECG between consecutive R waves, representing the ventricular rate (PR) interval, and QTc interval with Fridericia's correction method (QTcF) and QTc interval with Bazett's correction method (QTcB) were measured. Number of participants with clinically significant abnormal ECG findings were reported. Clinical significance was determined by the investigator.
Time Frame: Up to approximately 2.1 months
Population: as for outcome 8
Measure: Count of Participants; unit: Participants
Arm/Group | All Participants | ASN51 Low Dose | ASN51 Medium Dose | ASN51 High Dose
Number analyzed (Participants) | 3 | 3 | 1 | 1
Participants | 0 | 0 | 0 | 0

13. Secondary Outcome: Number of Participants With Clinically Significant Abnormal Physical Examinations
Description: Complete physical examination including general appearance; head, eyes, ears, nose, and throat; and cardiovascular, dermatologic, respiratory, gastrointestinal, musculoskeletal, and neurologic systems were performed. Number of participants with clinically significant abnormal physical examinations were reported. Clinical significance was determined by the investigator.
Time Frame: Up to approximately 2.1 months
Population: as for outcome 8
Measure: Count of Participants; unit: Participants
Arm/Group | All Participants | ASN51 Low Dose | ASN51 Medium Dose | ASN51 High Dose
Number analyzed (Participants) | 3 | 3 | 1 | 1
Participants | 0 | 0 | 0 | 0

14. Secondary Outcome: Plasma Concentration of ASN51 at Each Post-dose PET Scan
Time Frame: 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, and 16 hours post-dose on Day 1; 24 and 36 hours post-dose on Day 2; 48 hours post-dose on Day 3 and 72 hours post-dose on Day 4
Population: PK analysis population included the participants who provided evaluable data for the comparisons of interest. The participants had at least one quantifiable plasma concentration. Number analyzed is the number of participants with data available for analysis at specified time points.
Measure: Mean (Standard Deviation); unit: nanograms/milliliter (ng/mL)
Arm/Group | ASN51 Low Dose | ASN51 Medium Dose | ASN51 High Dose
Number analyzed (Participants) | 3 | 1 | 1
nanograms/milliliter (ng/mL)
  Day 1: 0.5 hour post-dose | 37.0 (8.78) | 192.0 | 43.5
  Day 1: 1 hour post-dose | 93.0 (6.16) | 181.0 | 189.0
  Day 1: 1.5 hours post-dose | 90.0 (7.79) | 159.0 | 293.0
  Day 1: 2 hours post-dose | 87.1 (11.98) | 144.0 | 283.0
  Day 1: 3 hours post-dose | 83.6 (8.92) | 142.0 | 245.0
  Day 1: 4 hours post-dose | 80.5 (17.12) | 134.0 | 253.0
  Day 1: 6 hours post-dose | 66.2 (7.77) | 121.0 | 199.0
  Day 1: 8 hours post-dose | 66.9 (11.22) | 115.0 | 201.0
  Day 1: 12 hours post-dose | 59.9 (9.73) | 103.0 | 153.0
  Day 1: 16 hours post-dose | 45.0 (6.74) | 96.9 | 153.0
  Day 2: 24 hours post-dose | 45.5 (6.24) | 81.7 | 133.0
  Day 2: 36 hours post-dose | 34.1 (4.71) | 58.2 | 95.3
  Day 3: 48 hours post-dose | 30.4 (3.37) | 46.3 | 88.2
  Day 4: 72 hours post-dose | 20.5 (1.28) | 28.9 | 54.8

15. Secondary Outcome: Estimated O-GlcNAcase Receptor Occupancy (RO) by Plasma Concentration of ASN51 and PET Scan
Description: Occupancy estimates were plotted against plasma concentrations of ASN51, corresponding to the start of each post-dose PET scan. Participant wise data was reported for this outcome measure.
  Row titles include participant number, PET scan session, post-dose time, and plasma concentration.
Time Frame: At 6 hours post-dose on Day 1 (for participant 1) and 31 hours post-dose on Day 1 (for participants 2 and 3), and at 48 hours post-dose on Day 1 (all participants)
Population: PET population included participants who received the study medication, had a baseline PET scan, at least one post-baseline PET scan, and a PK result immediately preceding PET scan. No summary analysis was done due to low number of participants, therefore participant-wise data are reported. Here, "number analyzed" signifies specific participant evaluated in respective arm at a specified timepoint.
Measure: Number; unit: percentage of receptor occupancy
Arm/Group | ASN51 Low Dose | ASN51 Medium Dose | ASN51 High Dose
Number analyzed (Participants) | 3 | 1 | 1
percentage of receptor occupancy
  Participant 1: PET Scan 2, 6 hours at 199.0 ng/mL: number analyzed (Participants) | 0 | 0 | 1
  Participant 1: PET Scan 2, 6 hours at 199.0 ng/mL |  |  | 92.2
  Participant 1: PET Scan 3, 48 hours at 30.3 ng/mL: number analyzed (Participants) | 1 | 0 | 0
  Participant 1: PET Scan 3, 48 hours at 30.3 ng/mL | 68.2 |  |
  Participant 2: PET Scan 2, 31 hours at 42.2 ng/mL: number analyzed (Participants) | 1 | 0 | 0
  Participant 2: PET Scan 2, 31 hours at 42.2 ng/mL | 84.5 |  |
  Participant 2: PET Scan 3, 48 hours at 29.4 ng/mL: number analyzed (Participants) | 1 | 0 | 0
  Participant 2: PET Scan 3, 48 hours at 29.4 ng/mL | 79.4 |  |
  Participant 3: PET Scan 2, 31 hours at 65.8 ng/mL: number analyzed (Participants) | 0 | 1 | 0
  Participant 3: PET Scan 2, 31 hours at 65.8 ng/mL |  | 89.7 |
  Participant 3: PET Scan 3, 48 hours at 26.7 ng/mL: number analyzed (Participants) | 1 | 0 | 0
  Participant 3: PET Scan 3, 48 hours at 26.7 ng/mL | 75.9 |  |

16. Secondary Outcome: Receptor Occupancy as Assessed by Plasma Concentration That Corresponds to 50% Occupancy (EC50)
Description: Occupancy estimates were plotted against plasma concentrations of ASN51, corresponding to post-dose PET scan. The following model was fitted to occupancy data set: Occ=100*Cp/Cp+EC50. Where Occ was the target occupancy (%), Cp was measured plasma concentration of ASN51 (ng/ml) and EC50 was the plasma concentration of ASN51 that corresponds to 50% occupancy. The relationship between exposure and occupancy was explored by direct fitting of a saturation model to pooled (across participants and scans) VT data, to obtain an estimate of EC50 for occupancy by ASN51.
Time Frame: At 6, 31 and at 48 hours post-dose on Day 1
Population: PET population included participants who received the study medication, had a baseline PET scan, at least one post-baseline PET scan, and a PK result immediately preceding PET scan.
Measure: Mean (95% Confidence Interval); unit: ng/mL
Groups:
- All Participants: Participants received low, medium, and high doses of ASN51 (as assigned according to the protocol), orally on Day 1 of imaging sessions 2 and 3 before the PET scan during the study.
Arm/Group | All Participants
Number analyzed (Participants) | 3
ng/mL | 9.4 [6.4 to 12.3]

ADVERSE EVENTS:
Time Frame: Up to approximately 2.1 months
Description: Safety analysis set included participants from the all-treated set who had at least one safety assessment post-baseline.
Arm/Group | All Participants | ASN51 Low Dose | ASN51 Medium Dose | ASN51 High Dose
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/3 | 0/1 | 0/1
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/3 | 0/1 | 0/1
Other Adverse Events (participants affected / at risk) | 2/3 | 0/3 | 1/1 | 0/1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | All Participants (N=3) | ASN51 Low Dose (N=3) | ASN51 Medium Dose (N=1) | ASN51 High Dose (N=1)
Catheter site related reaction (General disorders) | 2 | 0 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Dysgeusia (Nervous system disorders) | 1 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Agreement finally allows PI to publish independently.

DOCUMENTS (2):
  • Study Protocol (2021-05-19): https://cdn.clinicaltrials.gov/large-docs/98/NCT06390098/Prot_000.pdf
  • Statistical Analysis Plan (2021-11-17): https://cdn.clinicaltrials.gov/large-docs/98/NCT06390098/SAP_001.pdf